CLINICAL TRIAL: NCT02664727
Title: Effects of Acute Exercise on Psychological, Physiological, Biochemical and Alcohol-related Parameters in Individuals With Alcohol Use Disorders
Brief Title: Effects of Acute Exercise on Various Parameters in Individuals With Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: European Social Fund (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Dr, University of Thessaly
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UThessaly
Record Dates: First submitted 2016-01-15; First posted 2016-01-27 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Heavy Drinking; Alcohol Abuse; Alcohol Dependence; Alcohol Use Disorder
Keywords: alcohol; alcohol abuse; alcohol dependence; alcohol use disorder; heavy drinking; alcohol abuse cessation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heavy drinkers (Experimental): The effects of acute exercise in heavy drinkers. Participants will cycle on ergometer for 30 min at 50-60% of Heart Rate Reserve (HRR).
  Interventions: Behavioral: The effects of acute exercise in heavy drinkers
- Alcoholic patients (Experimental): The effects of acute exercise in alcoholic patients. Participants will cycle on ergometer for 30 min at 55-60% of Heart Rate maximal (HRmax).
  Interventions: Behavioral: The effects of acute exercise in alcoholic patients

INTERVENTIONS:
Behavioral: The effects of acute exercise in heavy drinkers — A group of heavy drinkers and a group of healthy controls (individuals without alcohol use disorders) will cycle on a cycle ergometer for 30 min at 50-60% of HRR. Before and immediately after exercise blood will be drawn and psychological and physiological parameters will be measured.
  Arms: Heavy drinkers
Behavioral: The effects of acute exercise in alcoholic patients — A group of alcoholic patients (10-14 days after detoxification) and a group of healthy controls (individuals without alcohol use disorders) will cycle on a cycle ergometer for 30 min at 55-60% of HRmax. Before and immediately after exercise blood will be drawn and psychological and physiological parameters will be measured.
  Arms: Alcoholic patients

SUMMARY:
The purpose of this research is to examine the effects of exercise of different intensities on psychological, physiological, biochemical, physiological and alcohol-related parameters in individuals with alcohol use disorders (heavy drinkers and alcoholic patients) in order to investigate possible biochemical mechanisms by which exercise may be a healthy alternative to alcohol abuse. For that purpose, a control group of individuals that do not exceed the limits for moderate alcohol use will be included.

DETAILED DESCRIPTION:
The mechanism of incentives that lead people to unhealthy habits such as excessive alcohol consumption is not only social, personal, and psychological, but also associated with neurochemical and neurobiological mechanisms.

Several programs have been developed to stop excessive drinking, but the success rates are small, while the relapse rates are very high, reaching up to 90%. Although there is some evidence for the beneficial effects of exercise on alcohol use disorders (AUDs), research is limited. The present study investigates whether exercise could be a safe adjunct therapy for alcohol abuse cessation, and the possible mechanisms involved.

One of the basic assumptions is that the appropriate form of exercise in individuals with AUDs will contribute to the secretion of beta-endorphin, which in combination with psychological pleasure, vitality, change of mood, reduced stress, increased confidence, and the shift of attention will help people to follow healthy lifestyles and abhor alcohol.

The research project is divided in three phases. In the first phase, (current study) the effect of acute exercise in critical psychological, physiological, biochemical and alcohol-related parameters associated with excessive alcohol consumption will be examined. In the second phase, a long-term exercise program in conjunction with psychological support strategies aimed at alcohol abuse cessation will be developed, implemented and evaluated. Finally, in the third phase, based on the results of the previous phases, awareness programs in adolescent and adult populations will be designed and implemented as well as the dissemination of results and evaluation of the project will take place.

ELIGIBILITY:
For alcoholics:

Inclusion Criteria:

* Confirmed alcohol addiction according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria in the past, after detoxification phase, lack of dependence on other substances
* Alcohol Use Disorders Identification Test (AUDIT) score>20

Exclusion Criteria:

* Medical conditions or medication use that would preclude participation in aerobic exercise

For heavy drinkers:

Inclusion Criteria:

* Men drinking >14 drinks/week or >4 drinks/occasion; Women drinking >7 drinks/week or >4 drinks/occasion (1 drink = 14 grams of pure alcohol; definition of the National Institute on Alcohol Abuse and Alcoholism (NIAAA) for drinking at low risk for developing an AUD; NIAAA, 2014)
* Individuals drinking 5 or more drinks on the same occasion on each of 5 or more days in the past 30 days (1 drink = 14 grams of pure alcohol; definition of the Substance Abuse and Mental Health Services Administration for heavy drinking; NIAAA, 2014)
* AUDIT score>8

Exclusion Criteria:

* Medical conditions or medication use that would preclude participation in aerobic exercise

For healthy controls:

Inclusion Criteria:

* Men drinking <14 drinks/week or <4 drinks/occasion; Women drinking <7 drinks/week or <4 drinks/occasion (1 drink = 14 grams of pure alcohol; definition of the NIAAA for drinking at low risk for developing an AUD; NIAAA, 2014)
* Individuals drinking <5 drinks on the same occasion on each of 5 or more days in the past 30 days (1 drink = 14 grams of pure alcohol; definition of the Substance Abuse and Mental Health Services Administration for heavy drinking; NIAAA, 2014)
* AUDIT score<8

Exclusion Criteria:

* Medical conditions or medication use that would preclude participation in aerobic exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in Urge to drink score | Before (0 min) and after exercise trial (30 min)
  According to questionnaire
Changes in Beta-endorphin levels | Before (0 min) and after exercise trial (30 min)
  Measured by radioimmunoassay (RIA)
Changes in Cortisol levels | Before (0 min) and after exercise trial (30 min)
  Measured by radioimmunoassay (RIA)
Changes in Adrenocorticotrophic hormone (ACTH) levels | Before (0 min) and after exercise trial (30 min)
  Measured by radioimmunoassay (RIA)
Changes in Catecholamines (epinephrine, norepinephrine, dopamine) levels | Before (0 min) and after exercise trial (30 min)
  Measured by radioimmunoassay (RIA)
Changes in C-reactive protein (CRP) levels | Before (0 min) and after exercise trial (30 min)
  Semi-quantitative estimation with CRP Latex test kit
Changes in Complete blood count values | Before (0 min) and after exercise trial (30 min)
  Autoanalyzer
Changes in Lactic acid levels | Before (0 min) and after exercise trial (30 min)
  Measured using photometry
Changes in Erythrocyte sedimentation rate (ESR) values | Before (0 min) and after exercise trial (30 min)
  Wintrobe Method
Changes in γ-Glutamyltransferase (GGT) levels | Before (0 min) and after exercise trial (30 min)
  Measured with commercial kit
Changes in Aspartate Aminotransferase (AST) levels | Before (0 min) and after exercise trial (30 min)
  Measured with commercial kit
Changes in Alanine Aminotransferase (ALT) levels | Before (0 min) and after exercise trial (30 min)
  Measured with commercial kit

SECONDARY OUTCOMES:
Sit and reach flexibility test for the hamstrings muscles and lower back | Before trial (baseline)
  Each participant sits on the floor with legs stretched out straight ahead, reaches out and holds that position for at 1-2 seconds while the distance is recorded.
Grip strength | Before trial (baseline)
  Handgrip strength test
Number of push-ups performed in one minute | Before trial (baseline)
Number of sit-ups performed until exhaustion | Before trial (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Theodorakis, PhD, Study Chair — University of Thessaly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Georgakouli K, Manthou E, Fatouros IG, Deli CK, Spandidos DA, Tsatsakis AM, Kouretas D, Koutedakis Y, Theodorakis Y, Jamurtas AZ. Effects of acute exercise on liver function and blood redox status in heavy drinkers. Exp Ther Med. 2015 Dec;10(6):2015-2022. doi: 10.3892/etm.2015.2792. Epub 2015 Oct 13. PMID 26668589